CLINICAL TRIAL: NCT02349893
Title: Radiofrequency Ablation for Multi-level Obstructive Sleep Apnea: A Single-arm, Multicenter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Surgical Technologies Europe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2015-01-24; First posted 2015-01-29 (Estimated); Results first posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Apnea, Sleep
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RFA treatment (Experimental): RFA treatment performed with CelonProSleep plus device
  Interventions: Device: RFA treatment

INTERVENTIONS:
Device: RFA treatment — RFA treatment using CelonProSleep plus system

SUMMARY:
The United States is currently experiencing an increase in the incidence and prevalence of obstructive sleep apnea (OSA). With prevalence in middle-aged adults of 2 to 4% of the population, untreated OSA has been implicated in increased risk for cardiovascular disease, including hypertension and heart failure, daytime sleepiness, and increased risk of motor vehicle accidents.

This study was design in order to evaluate the CelonProSleep plus for multi-level radiofrequency ablation (RFA) of the palate and base of tongue as a treatment for mild to moderate obstructive sleep apnea syndrome (OSAS).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 22 years)
* Self-report of daytime somnolence
* Body mass index (BMI) ≤ 32
* Mild to moderate obstructive sleep apnea (AHI 10 - 30; lowest O2 sat ≥ 80%)
* Evidence of palate and tongue base collapse on supine fiberoptic examination
* Non-compliant with or refusal of continuous positive airway pressure therapy (CPAP) (< 4 hours per night by patient report)
* No prior surgical treatment for OSAS other than nasal surgery
* Willing and capable of providing informed consent

Exclusion Criteria:

* Another significant sleep disorder (e.g., insomnia, periodic limb movement)
* Tonsillar hypertrophy
* Chronic Obstructive Pulmonary Disease (COPD)
* Interstitial Lung Disease (ILD)
* Cystic Fibrosis
* Acute Repiratory Distress Syndrome (ARDS)
* Nasal or supraglottic obstruction on fiberoptic examination
* American Society of Anesthesiologists (ASA) class III ,IV, V
* Latex allergy
* Lidocaine allergy
* Pregnancy or plans to become pregnant Note: women of childbearing potential must demonstrate a negative pregnancy test upon enrollment; those patients qualified to progress to RFA must also demonstrate a negative pregnancy test within 7 days prior to the date of RFA procedure.
* Major depression or non-stabilized psychiatric disorder
* Drug or alcohol abuse
* Previous palatal or tongue surgery
* Stable or unstable angina
* congestive heart failure (CHF)
* moderate or severe valvular disease
* transient ischemic attack (TIA)/cardiovascular accident (CVA)
* Carotid stenosis or endarterectomy
* Anemia
* Room air oxygen saturation (SpO2) < 95%
* Pulmonary hypertension
* Dialysis
* Central or mixed apnea ≥ 10% of respiratory events
* Participation in another clinical study (enrolled in any concurrent study) whose investigational plan is judged to interfere or affect any of the measures of this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Nguyen, MD, Principal Investigator — Medical University of South Carolina
Locations (6):
- United States (6):
  - Alessi Clinic, Beverly Hills, California
  - Otolaryngology Colorado, Greenwood Village, Colorado
  - ENT of Georgia, Atlanta, Georgia
  - Bluesleep clinic, New York, New York
  - Institutional Review Board for Human Research (IRB), Charleston, South Carolina
  - Methodist Healthcare Foundation, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- RFA Treatment: RFA treatment performed with Celon ProSleep plus device, three treatment sessions of RF ablation of the soft palate (7 lesions) and the base of tongue (6 lesions)
Period: Overall Study
Arm/Group | RFA Treatment
Started | 56
Completed | 43
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | RFA Treatment
Number analyzed (Participants) | 56
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Results are presented separately for study completers (n=43) and study dropouts (n=13). The overall number of baseline participants is n=56 including all study completers and study dropouts.
  years
    Study completers: number analyzed (Participants) | 43
    Study completers | 50.67 (11.20)
    Study dropouts: number analyzed (Participants) | 13
    Study dropouts | 53.75 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Results are presented separately for study completers (n=43) and study dropouts (n=13). The overall number of baseline participants is n=56 including all study completers and study dropouts.
  Participants
    Study completers: number analyzed (Participants) | 43
    Study completers: Female | 13
    Study completers: Male | 30
    Study dropouts: number analyzed (Participants) | 13
    Study dropouts: Female | 2
    Study dropouts: Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 44
  More than one race | 0
  Unknown or Not Reported | 8
Apnea Hypopnea Index [Mean (Standard Deviation); unit: No. of apneas/hypopneas per h of sleep] — Population: Results are presented separately for study completers (n=43) and study dropouts (n=13). The overall number of baseline participants is n=56 including all study completers and study dropouts.
  No. of apneas/hypopneas per h of sleep
    Study completers: number analyzed (Participants) | 43
    Study completers | 19.70 (7.10)
    Study dropouts: number analyzed (Participants) | 13
    Study dropouts | 19.15 (6.93)

OUTCOME MEASURES:

1. Primary Outcome: Mean Apnea Hypopnea Index (AHI) at 6 Months Post-baseline
Description: The primary endpoint is the apnea hypopnea index (AHI) at 6 months post-baseline.
Time Frame: 6 months following last treatment
Population: The apnea hypopnea index after the treatment was analyzed for all study completers.
Measure: Mean (Standard Deviation); unit: No. of apneas/hypopneas per h of sleep
Arm/Group | RFA Treatment
Number analyzed (Participants) | 43
No. of apneas/hypopneas per h of sleep | 9.86 (8.28)

ADVERSE EVENTS:
Time Frame: Adverse Events were documented from first RFA treatment until the final follow-up visit after 6 months
Arm/Group | RFA Treatment
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

LIMITATIONS AND CAVEATS:
This was a multicenter single-arm study. Further randomized controlled trails are needed to obtain higher level of evidence.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT02349893/Prot_SAP_000.pdf